CLINICAL TRIAL: NCT01623427
Title: The AVATAR Trial: Applying VAcuum To Accomplish Reduced Wound Infections in Laparoscopic Pediatric Surgery
Brief Title: The AVATAR Trial: Applying VAcuum To Accomplish Reduced Wound Infections
Acronym: AVATAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting enough patients
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Richard Keijzer, assistant professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2012:037
Record Dates: First submitted 2012-06-11; First posted 2012-06-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Post-laparoscopy Umbilical Port-site Wound Infection
Keywords: pediatric; laparoscopy; vacuum; dressing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vacuum (Experimental): the group of patients assigned to application of vacuum to the wound dressing
  Interventions: Procedure: Application of vacuum
- Control (Active Comparator): The dressing for the umbilical port site will be the same as the experimental group, except for the application of vacuum. The control group will have no vacuum applied to the wound dressing.
  Interventions: Procedure: No vacuum

INTERVENTIONS:
Procedure: Application of vacuum — The vacuum will be applied to the wound dressing of the umbilical port site using a 22 g needle on a 10 ml syringe passed percutaneously from the outside of the dressing into the gauze and the air around the gauze is evacuated.
  Other Names: Non applicable
  Arms: Vacuum
Procedure: No vacuum — Except for the vacuum, the wound dressing for the umbilical port site will be the same. No vacuum will be applied to the wound dressing of this group
  Other Names: Non applicable
  Arms: Control

SUMMARY:
Postoperative pain and time taken to return to normal activities after laparoscopic surgery are significantly shorter. Wound infections still occur and contribute to prolonged hospital stays and morbidity. Typically, port incision sites are covered with a standard dressing (approximating strips and a gauze). Although the umbilical wound infection rate in laparoscopic surgery is considered to be low, a recent study by Muensterer and Keijzer showed that the umbilical wound infection rate after single incision laparoscopic appendectomy in children is approximately 7%. In the same retrospective study, the investigators demonstrated that a simple low cost vacuum dressing can significantly reduce the infection rate. The aim of this prospective randomized controlled trial is to determine if the simple vacuum dressing is superior to a standard dressing in reducing laparoscopic postoperative umbilical wound infections. All patients under 17 years of age undergoing a laparoscopic operation in the Children's Hospital will be randomized to a standard postoperative dressing or a standard postoperative dressing with vacuum applied to it. The vacuum will be applied with a 22g needle on a 10ml syringe passed percutaneously from outside the dressing into the gauze and the air around the gauze is evacuated. The umbilical wounds will be evaluated 8-10 days postoperatively in the clinical research unit of the Manitoba Institute of Child Heath according to a standardized and validated wound evaluation tool from the Canadian Center for Disease Control. Primary outcome measure in this study is postoperative wound infection. A sample size calculation using the retrospective data demonstrated that the investigators need 275 patients in each group for the Chi-squared test to have an 80% chance of detecting a difference in wound infection rate of 6% at the 5% level of significance. Based on the annual number of laparoscopic operations in the Children's Hospital (around 400) the investigators anticipate completing the inclusion of patients within a two-year period.

DETAILED DESCRIPTION:
The AVATAR Trial: Protocol

Applying VAcuum To Accomplish Reduced wound infections in laparoscopic pediatric surgery

Surgical Site Infections (SSIs) are the most common complication of surgery worldwide and one of the leading causes of morbidity and mortality in surgical patients. Literature has shown that patients who develop an SSI are five times more likely to require readmission to hospital within 30 days, 60% more likely to require ICU admission, and twice as likely to die. SSIs also carry a significant financial burden to the healthcare system. Annually in the US, SSIs account for over 900 million dollars spent in-hospital and $1.6 billion overall in health care. The average risk of developing an SSI from any surgical procedure is 1-4%. A landmark study by Horan, et al. in 1992 defined SSIs as any infection occurring within 30 days of an operation or up to 1 year if an implanted device was used. Infections were further classified as: superficial incisional, deep incisional, or organ/space, with diagnostic criteria on physical exam to support each category. This criterion for SSI diagnosis has since become the standard definition at the American Center for Disease Control (CDC) and worldwide.

Table 1: CDC Definition of an SSI.

Superficial Incisional SSI:

* Infection occurring within 30 days of an operative procedure AND
* Involves only skin or subcutaneous tissue of the incision AND
* Patient has at least 1 of the following:
* Purulent drainage from the superficial incision
* Organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision
* At least one of the following signs or symptoms: pain or tenderness; localized swelling, redness, or heat; superficial incision is opened by a surgeon and is culture-positive or not cultured. A culture negative finding does not meet this criterion.
* Diagnosis of a superficial incisional SSI by a surgeon

Deep Incisional SSI:

* Infection occurring within 30 days of an operative procedure if no implant OR within 1 year if an implant is used AND the infection appears to be related to the operative procedure AND
* Involves deep soft tissues (eg. fascial and muscle layers) of the incision AND
* Patients has at least one of the following:
* Purulent drainage from the deep incision but not from the organ/space component of the surgical site
* A deep incision spontaneously dehisces or is deliberately opened by a surgeon and is culture positive or not cultured when the patient has at least one of the following signs or symptoms: fever > 38 degrees Celsius or localized pain or tenderness. A culture negative does not meet this criterion.
* An abscess or other evidence of infection involving the deep incision is found on direct examination, during reoperation, or by histopathologic or radiologic examination.
* Diagnosis of a deep incisional SSI by a surgeon

Organ/Space SSI:

* Infection occurs within 30 days of an operative procedure if no implant was used OR within 1 year if an implant was used AND the infection appears to be related to the operative procedure AND
* Infection involves any part of the body (excluding the skin incision, fascia, or muscle layers) that is opened or manipulated during the operative procedure AND
* Patient has at least 1 of the following:
* Purulent drainage from a drain that is placed through a stab wound into the organ/space
* Organisms isolated from an aseptically obtained culture of fluid or tissue in the organ / space
* An abscess or other evidence of infection involving the organ / space that is found on direct examination, during reoperation, or by histopathologic or radiologic examination
* Diagnosis of an organ/space infection by a surgeon

Significant research has been undertaken to determine risk factors, prevention, and treatment of SSIs. Risk factors can generally be divided into procedure- and patient-specific risks. Horan, et al. grouped procedures into 4 wound classifications: clean, clean-contaminated, contaminated, and dirty. They found that clean operations carried an average risk of 1% while dirty surgeries carried a risk > 27%. Other procedure-specific risk factors that have been identified include: length of the procedure, degree of hemostasis, tissue trauma, and use of drains. Patient-specific risk factors include: age, smoking, obesity, diabetes, poor nutrition, and compromise of the immune system.

While there is a large body of research addressing SSIs in adults, very few papers have addressed the development of SSIs in the pediatric population. Bucher, et al. found that SSI prediction models used in adults are not generalizable to pediatrics. Extremes of age, immune naivety, general physiology, and indications and types of procedures undertaken on children are significantly different than those faced by adults. Research has found that procedure-specific risks are much more heavily weighted in pediatric populations than patient-specific risks.

A number of interventions have aimed at reducing procedure-specific risk factors, including: clipping rather than shaving hair, chlorhexidine vs iodine skin preparation, steri-strips vs sutures vs tissue glue for closure, and the use of prophylactic antibiotics. However, very few studies have looked at post-operative dressings as a role player in reducing SSIs. A recent Cochrane Review on this subject revealed that there is currently no evidence to suggest that any dressing significantly reduces the risk of SSI in wounds healing from primary intention. However, the Cochrane review also revealed that the 16 randomized controlled studies included in the review were generally of poor quality, small sample size, and/or high bias. Cochrane listed the following aspects as attributes of an ideal dressing:

* ability to absorb and contain exudate without leakage
* lack of particulate contaminants left in wound by dressing
* thermal insulation
* impermeability to water and bacteria
* ability to use with different types of skin closure (ie. stapes, sutures)
* avoidance of wound trauma on removal
* minimal frequency of dressing changes
* provision of pain relief
* cosmesis and comfort
* effect on formation of scar tissue

In 2011, the investigators published a pilot study that showed that a simple, cost-effective vacuum dressing could reduce wound infection rates in pediatric laparoscopic appendectomies by 6%. This dressing is fashioned by placing a sterile 2 by 2 inch gauze over the umbilical port site and covering it with a bioocclusive dressing, such as an op-site. A 22-gauge needle is then inserted subcutaneously to remove air from the dressing, thereby creating a vacuum atmosphere. This dressing fulfills all the criteria from the Cochrane review of preferred attributes, is easy to apply, and inexpensive.

The use of negative-pressure wound treatments (NPWT) is not a novel concept - however, specialized VAC dressings are costly (at approx $107/day) and generally reserved for complex, debilitating wounds. NPWT are thought to promote wound healing by removing local edema, improving vascular and lymphatic flow, decreasing bacterial density, and promoting angiogenesis and formation of granulation tissue. Minimal literature is available on the utility of these dressings in children. Six studies that have shown NPWT to be effective in healing complex wound dehiscence in the pediatric population; however, to the investigators' knowledge, no study has yet been undertaken to look at the role of NPWT in SSI prevention and healing of non-complex wounds in either pediatrics or adults.

The aim of this study is to address this very issue by undertaking a randomized controlled trial with sufficient statistical power to prove (or disprove) that a simple, vacuum dressing can be effective at reducing the SSI rate in children undergoing any laparoscopic procedure.

The primary outcome measure in this study is the rate of postoperative wound infection at the umbilical port site. A sample size calculation using the pilot study data demonstrated that the investigators need 275 patients in each group for the Chi-squared test to have an 80% chance of detecting a difference in wound infection rate of 6% with a 5% level of significance. Approximately 600 patients will need to be recruited from the Children's Hospital to ensure sufficient statistical power. Based on the annual number of laparoscopic procedures in the Children's Hospital (approximately 400) the investigators anticipate completing the inclusion of patients within a two-year period. Candidates will be screened for eligibility upon booking operative time for a laparoscopic surgery. These surgeries may be either elective or emergent in nature. Patients will be recruited by the pediatric surgery service that will meet with the patients and their parents/guardians prior to the operation to discuss the purpose of the trial and their role, should they choose to participate. Written information will be supplied and consent will be obtained from the patient directly or their parent/guardian by the nurse in clinic or the operating room. Once enrolled, patients will be randomized to one of two arms: one group will receive a simple vacuum dressing to their umbilical port (experimental) while the other group will receive the standard dressing without vacuum (control). Randomization will take place after the operation has been completed and will be done via a computer-generated list of numbers in a 1:1 ratio using the online tool Research Randomizer.

All patients will be prepped with chlorhexidine and draped using sterile paper drapes. The umbilical incisions will be made in a horizontal manner and the trochar will be introduced using the Hasson technique.

Both groups will undergo fascial closure of the umbilical wound with a figure-of-8, 0 vicryl stitch and subsequent umbilical port closure with 5-0 biosyn simple interrupted subcutaneous sutures. A 2x2 sterile gauze will be applied with a simple bio-occlusive dressing (ie. op-site). In the vacuum dressing group, a 22-gauge needle will be introduced subcutaneously into the dressing and air will be suctioned out using a 10 cc syringe.

Post-operatively, the dressings in both groups will be removed after 48 hrs, either by the patients (or their parents) if the patient is discharged home or the house staff on the ward if they are an inpatient.

An independent nurse from the clinical research unit at the Manitoba Institute of Child Health (MICH) who is blinded to the treatment groups will examine the patients at 8-10 days post-operatively and diagnose any surgical site infections using the criteria provided by the CDC. Funding for the MICH nurse has already been approved (see budget). The timeframe for follow up was chosen because it will minimize the likelihood of patients being lost to follow up while maximizing the opportunity for detection of infection, since the majority of SSIs are apparent by postoperative day 3-5.

Based on the pilot study, it is unlikely that the simple vacuum dressing will increase the rates of SSI however as the data is accrued the investigators will assess the results in real time for a disparity in SSIs greater than 10% between the study and experimental groups. Should this disparity exist, in either direction, recruitment will temporarily be held while the results are analyzed for their statistical significance at that point. If the results are significant, the investigators will consider terminating the trial before all 600 patients are recruited and changing practice accordingly.

Data collected from the trial will be stored on a computer kept in a secure location on the Health Sciences campus. The file will be kept for a period of 25 years (or when the youngest child in the study turns 25). Only members of the research group will have access to the password-protected server where the data is kept. As patients are recruited, they will be assigned a unique identification number that is separate from their PHIN or hospital ID. This number will be used to organize the data instead of the patient's name or health information. Only the patient's date of birth, weight, sex, diagnosis, procedure type and duration, estimated blood loss, length of stay, and presence or absence of SSI will be recorded. Since identifying information about the patients will not be recorded, the investigators will not directly contact the patients with the results of the trial. Instead, patients will be provided with an email address (avatar.clinical.trial@gmail.com that they can contact, from which the investigators will periodically send out updates about the trial.

ELIGIBILITY:
Inclusion Criteria:

* age 0-17 years old
* any emergency or elective laparoscopic procedure requiring an umbilical port

Exclusion Criteria:

* immunocompromise (acquired or iatrogenic)
* malignancy
* requiring blood transfusion within 6 weeks of surgery
* history of splenectomy
* significant comorbid conditions, such as severe cardiopulmonary disease
* presence of any chronic abdominal wound, cellulitis, or enterocutaneous fistula
* pregnancy
* smoker
* BMI > 30
* inability to attend follow up
* language barrier

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The rate of postoperative wound infections at the umbilical port site. | prospective
  The primary outcome measure: postoperative wound infection at the umbilical port site will be blindly evaluated at 8-10 days postoperatively according to the criteria provided by the CDC by an independent nurse from the clinical research unit at the Manitoba Institute of Child Health (MICH) The timeframe for follow up was chosen because it will minimize the likelihood of patients being lost to follow up while maximizing the opportunity for detection of infection, since the majority of SSIs are apparent by postoperative day 3-5.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Keijzer, MD PhD MSc, Principal Investigator — University of Manitoba; Robin Visser, MD, Study Director — University of Manitoba
Locations (1):
- Children's Hospital of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Muensterer OJ, Keijzer R. A simple vacuum dressing reduces the wound infection rate of single-incision pediatric endosurgical appendectomy. JSLS. 2011 Apr-Jun;15(2):147-50. doi: 10.4293/108680811X13071180406592. PMID 21902964